CLINICAL TRIAL: NCT01565226
Title: Capnography in Neonates Ventilated With High Frequency Ventilation: Prospective, Observational Multi-Center Study
Status: Completed | Type: Observational
Sponsor: Oridion (Industry)
Responsible Party: Sponsor
Organization: Medtronic - MITG (Industry)
Other Study IDs: D007171
Record Dates: First submitted 2012-03-25; First posted 2012-03-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Intubated Neonates That Require High Frequency Ventilation
Keywords: Capnography; CO2; neonates; High Frequency ventilation (HFV)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Open: open, observational study

SUMMARY:
* This will be an observational study. Respiratory data will be recorded using Capnostream20p. There will be no use in the recorded data for the medical care of the patients. Other clinical data will be captured in the CRF. Similar study is currently conducted in Bnai Zion MC since 2008. Thirty four (34) patients have been recruited without any adverse events.
* During the study the medical team will capture in the CRF the following: Blood gas and distal capnography values at time of sampling, ventilator settings at time of sampling.
* Changes made in the ventilation parameters, blood gas time and results, concomitant treatment (e.g. suction) and concomitant medication (respiratory related e.g. surfactant), vital signs all these will be retrieved from the patient's medical charts.

ELIGIBILITY:
Inclusion Criteria:

* Intubated neonates with double-lumen ETT (Uncuffed Tracheal Tube, Mallinckrodt Inc., Chih, Mexico)
* Neonates that their respiratory condition requires HFV
* Neonates expected to have at least 3 pairs of distal capnography measurements and blood gas samplings.

Exclusion Criteria:

* Intubated neonates with single-lumen ETTs
* Neonates who are ventilated with conventional ventilation
* Any significant medical condition which, at the investigator's discretion, may interfere with the study.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neonates
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of measuring distal capnography on HFV and to assess its correlation and agreement with PaCO2 in infants ventilated with HFV in a prospective study. | August 2012 - February 2015

CONTACTS AND LOCATIONS:
Overall Officials: Amir Kugelman, Prof., Principal Investigator — Bnai Zion MC, Haifa Israel
Locations (3):
- Israel (3):
  - Soroka MC, Beersheba
  - Bnai Zion MC, Haifa
  - Shaare Zedek MC, Jerusalem